CLINICAL TRIAL: NCT07065825
Title: A Retro-Prospective Observational Study on Causes, Characteristics, Intraoperative Management and Impact on Prognosis
Brief Title: Tumor Rupture During Robotic Partial Nephrectomy
Acronym: RUPTURE
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: Fundación Investigación Hospital IMED Valencia, Valencia, Spain (Unknown); Hospital Clinic de Barcelona, Barcelona, Spain (Unknown); The Cleveland Clinic (Other); Fundacio Puigvert (Other); San Raffaele University Hospital, Italy (Other); Guy's and St Thomas' NHS Foundation Trust (Other); University Hospital, Bordeaux (Other); Fox Chase Cancer Center (Other); ASST Grande Ospedale Metropolitano Niguarda (Other); Azienda Ospedaliero-Universitaria Careggi (Other); Ospedale San Luigi Gonzaga, Orbassano (Unknown); Changhai hospital of Navy Medical University (Unknown); St. George's Hospital, London (Other); Frimley Health NHS Foundation Trust (Unknown); Icahn School of Medicine at Mount Sinai (Other); Rennes University Hospital (Other); University of Illinois at Chicago (Other); University of California, San Diego (Other); Hospital da Luz, Lisboa (Unknown); Swedish Medical Center (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); St. Antonius Hospital Gronau (Other); Regina Elena Cancer Institute (Other); Pitié-Salpêtrière Hospital (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Onze Lieve Vrouwziekenhuis Aalst (Other); Hannover Medical School (Other); Royal Free and University College Medical School (Other); Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other); Memorial Sloan Kettering Cancer Center (Other); The Netherlands Cancer Institute (Other); A.O.U. Città della Salute e della Scienza - Molinette Hospital (Other); University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: 674CET
Record Dates: First submitted 2025-07-02; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Kidney Cancer; Renal Neoplasms
Keywords: robotic; robotic surgery; partial nephrectomy; tumor rupture; tumour rupture; tumor resection; kidney cancer; small renal mass; robotic partial nephrectomy; robot-assisted partial nephrectomy
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who experienced tumor rupture during robotic partial nephrectomy: Patients who experienced tumor rupture during RAPN (referred to an unintended breach of the tumor capsule with or without spillage of malignant tissue during tumor resection)
  Interventions: Procedure: robot-assisted partial nephrectomy

INTERVENTIONS:
Procedure: robot-assisted partial nephrectomy — Robotic-Assisted Partial Nephrectomy (RAPN) is a minimally invasive surgical procedure performed with the help of a robotic system to remove a kidney tumor while preserving as much healthy kidney tissue as possible. It is commonly used to treat small to medium-sized kidney tumors. Thanks to the precision of robotic technology, RAPN offers faster recovery, less postoperative pain, and fewer complications compared to traditional open surgery.
  Other Names: robotic partial nephrectomy; RAPN; RPN

SUMMARY:
The RUPTURE Project is a multi-center observational study aiming to understand tumor rupture during robotic partial nephrectomy (RAPN), a minimally invasive surgery used to treat kidney tumors. Tumor rupture-an unintended break of the tumor capsule during surgery-occurs in about 10-15% of cases but is poorly studied. This event may increase the risk of cancer recurrence or spread, but its true impact is still unclear.

The study includes adult patients who experienced a tumor rupture during RAPN. Researchers will collect data on patient and tumor characteristics, surgical techniques, how the rupture occurred and was managed, and long-term outcomes. Follow-up visits will monitor for recurrence, metastases, and survival for up to five years. No experimental treatments or extra procedures are involved; only standard care is followed.

By analyzing at least 100 cases from various hospitals, the study hopes to clarify whether tumor rupture affects prognosis and to identify risk factors and best practices for managing it. This could help improve patient safety, surgical strategies, and future clinical guidelines. All data are handled confidentially, and participation is voluntary.

DETAILED DESCRIPTION:
Background Robotic-assisted partial nephrectomy (RAPN) is a common, minimally invasive surgery used to remove kidney tumors while preserving healthy kidney tissue. While generally safe and effective, a complication called tumor rupture may occasionally occur. This means the tumor capsule (its outer layer) breaks during surgery, sometimes causing cancer cells to spill into the body. Although reported in up to 15% of surgeries, tumor rupture is not well understood, and its impact on long-term cancer outcomes remains unclear.

Purpose of the Study

This study, called the RUPTURE Project, aims to better understand tumor rupture during RAPN by answering key questions:

Does tumor rupture affect cancer recurrence or survival?

What causes it?

How can it be effectively managed during surgery?

How the Study Works This is a retro-prospective observational study, meaning it collects and analyzes both past and future cases of tumor rupture during RAPN. It involves multiple hospitals and surgical centers.

Who Can Participate? The study includes adult patients (18-80 years) who experienced a tumor rupture during RAPN and agree to participate. It excludes patients who had a radical nephrectomy (complete kidney removal), underwent open or laparoscopic surgery instead of robotic surgery, or had other complex medical conditions affecting the kidneys.

What Data Is Collected?

No additional procedures are required beyond standard clinical care. The study gathers information about:

Patient characteristics (age, health status, kidney function)

Tumor characteristics (size, location, type)

Surgical details (how the rupture occurred, surgical tools used, and how the situation was managed)

Pathological analysis (tumor grade, stage, margins)

Follow-up outcomes, including:

Local recurrence of the tumor

Spread (metastasis) to other parts of the body

Cancer-related and all-cause survival over a 5-year period

Why This Study Matters

Currently, there are no standardized guidelines for managing tumor rupture during kidney surgery. The RUPTURE Project will provide essential information to help:

Predict when and why ruptures occur

Guide surgeons on best practices during rupture events

Understand the long-term impact on patient health

Impact on Patients and Health Providers

The results of this study could lead to:

Safer surgeries with fewer complications

Improved guidelines for managing tumor rupture

Better information for patients facing kidney surgery

Potential changes in how surgeons plan and respond to complications

Study Duration The study will collect data over 2 years and follow up with patients for at least 5 years. A total of 100 or more cases of tumor rupture are expected to be analyzed across multiple centers.

Ethical and Privacy Considerations Participation is voluntary, and all patient data is handled confidentially, in compliance with European and Italian privacy laws (GDPR and national regulations). No experimental treatments or changes to care are made-this is strictly an observational study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who experienced tumor rupture during RAPN (referred to an unintended breach of the tumor capsule with or without spillage of malignant tissue during tumor resection)
* Patients who provide informed consent to participate
* Patients from 18 to 80 years of age.

Exclusion Criteria:

* Patients undergoing radical nephrectomy or other nephron-sparing procedures.
* Patients undergoing partial nephrectomy with other approaches (open, pure laparoscopic)
* Patients with multiple ipsilateral tumors
* Patients diagnosed with genetic abnormalities that increase the likelihood of developing renal cell carcinoma.
* Patients who deny consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of interest comprises all patients undergoing RAPN for renal mass.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
cumulative incidence of recurrences | From date of enrolment until the date of first documented event, assessed up to 60 months
  cumulative incidence of tumor local recurrences (at surgery site)
Cumulative incidence of Metastases | From date of enrolment until the date of first documented event, assessed up to 60 months
  cumulative incidence of tumor distant metastases
Cumulative incidence of Cancer-related Deaths | From date of enrolment until the date of first documented event, assessed up to 60 months
  Cumulative incidence of cancer-related deaths (deaths due to the disease). This will be evaluated through cancer-specific survival (CSS)
Cumulative incidence of All-cause Deaths | From date of enrolment until the date of first documented event, assessed up to 60 months
  Cumulative incidence of non-cancer-related deaths (deaths due to other cause) disease). This will be evaluated through overall survival (OS)

SECONDARY OUTCOMES:
Timing of tumor rupture | During surgery
  To evaluate the timing of tumor rupture (if it occurs during tumor isolation, at the early of tumor resection, almost at completion of the resection, at tumor grabbing for bagging).
type of tumor rupture | During surgery
  Will evaluate the type of rupture, focal vs. gross; with vs. without spillage of tumor cells
Cause of rupture | During surgery
  Will evaluate the cause of rupture (if it is due to the surgeon's move vs. an assistant's action)
Surgical instrument causing the rupture | During surgery
  Will evaluate which robotic instruments, or which assistant's instrument did cause the tumor rupture

OTHER OUTCOMES:
Tumor rupture Management Strategy 1 | During surgery
  Use of suction or other methods for controlling spillage: bagging vs. grasping
Tumor rupture Management Strategy 2 | During surgery
  CO2 insufflation pressure adjustments during rupture: Yes vs. No
Tumor rupture Management Strategy 3 | During surgery
  Conversion to open surgery after tumor rupture: yes vs. no
Tumor rupture Management Strategy 4 | During surgery
  Conversion to radical nephrectomy after tumor rupture: Yes vs. No.

CONTACTS AND LOCATIONS:
Locations (1):
- AOUI Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu P, Zhang S, Cao B, Huang J, Li Y, Cheng J, Lin W, Cheng J, Chen W, Zhu Y, Jiang S, Hu X, Guo J, Wang H. Does intraoperative cyst rupture of malignant cystic renal masses really have no negative impact on oncologic outcomes? World J Surg Oncol. 2022 Nov 25;20(1):369. doi: 10.1186/s12957-022-02824-7. PMID 36434718
- [Background] Bertolo R, Campi R, Amparore D; European Association of Urology (EAU) Young Academic Urologists (YAU) Renal Cancer Working Group. YAU renal cancer SPOTLIGHT: the understated challenge of tumor rupture during robotic partial nephrectomy. Minerva Urol Nephrol. 2025 Jun;77(3):417-421. doi: 10.23736/S2724-6051.25.06509-7. No abstract available. PMID 40528779